CLINICAL TRIAL: NCT03137550
Title: Combined Use of Multiple Biomarkers With Stress Testing to Detect Coronary Artery Disease
Acronym: COMBAT-CAD
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4023
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Main aim of the COMBAT-CAD-Study is to clarify, if the combination of stress testing with biomarkers improves the diagnostic accuracy.

Hypothesis of our study is that diagnosis of CAD can be improved by adding biomarkers to solely stress testing for the workup of patients with suspected CAD or progress of already known CAD.

DETAILED DESCRIPTION:
The COMBAT-CAD Study is an observational study with the aim to improve the diagnostic accuracy by a combination of stress testing with sensitive and specific biomarkers in detecting coronary artery disease or its progress. The main subjects are all patients with CAD or suspicion of CAD sent to the University Heart Center Hamburg. In these patients, ECG, laboratory examination, symptoms or transthoracic echocardiography in rest could not rule out CAD or progress of known CAD. The hypothesis of the study is that detection of CAD can be improved by adding biomarkers to stress testing for the diagnostic workup of patients with suspected CAD or progress of already known CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Every patient referred to coronary angiography, or diagnostic work-up with suspicion of CAD or progress of CAD (in case of CABG patients or already treated with PCI)

Exclusion Criteria:

1. Insufficient knowledge of the German language (able to understand and write the German language)
2. Physical or psychological incapability to take part in the investigation
3. Persons with no sufficient language ability in German to understand the provided study information material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible are all patients who receive stress testing ordered by a physician of the University Heart Center and who are willing and able to participate in an observational study. Participants of interest are outpatients and inpatients of the University Heart Centre.
Sampling Method: Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of coronary artery disease | Within the initial diagnostic evaluation process (maximum within 30 days)
  The diagnosis of coronary artery disease through stress testing alone and combined with cardiac biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, MD, Principal Investigator — Head of the Department
Locations (1):
- Department of General and Interventional Cardiology, University Heart Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No